CLINICAL TRIAL: NCT00696358
Title: Comparative Study of 308nm Excimer Lamp and 308nm Excimer Laser in the Treatment of Vitiligo
Brief Title: Excimer Lamp Versus Excimer Laser in Vitiligo Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Other Study IDs: NICE-VIT1
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Vitiligo
Keywords: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Lasers, Excimer

ARMS (2):
- A (Active Comparator): 308 nm excimer lamp
  Interventions: Radiation: 308nm excimer lamp
- B (Active Comparator): 308 nm excimer laser
  Interventions: Radiation: 308nm excimer laser

INTERVENTIONS:
Radiation: 308nm excimer lamp — 50 mJ/cm² below the MED (minimal erythemal dose) and progressive increase Twice a week for 12 weeks
  Arms: A
Radiation: 308nm excimer laser — 50 mJ/cm² below the MED (minimal erythemal dose) and progressive increase Twice a week for 12 weeks (same doses will be used between the 2 arms)
  Arms: B

SUMMARY:
308 nm excimer lamp and 308 nm excimer laser have both provide interesting results in treating vitiligo. They have the same wavelength but the type of emission of the photons is different. To date there is no direct comparative data concerning these two devices in this indication.

The aim of the study is to make an intra-individual prospective comparison between these two phototherapies.

ELIGIBILITY:
Inclusion Criteria:

* patient above 18
* vitiligo for more than 3 months
* at least 2 vitiligo symmetric patches more than 10cm²
* to read and understand the inform consent
* to have a social security number
* non pregnant for women

Exclusion Criteria:

* pregnant women
* keloids
* history of radiotherapy or skin cancer in the treated areas
* treatment for vitiligo in the past 4 weeks
* phototherapy in the past 12 weeks; history of photodermatosis
* treatment inducing photosensibilization
* immunosuppression
* patient who participated in a study in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Repigmentation rate in the treated areas | 12 weeks

SECONDARY OUTCOMES:
Tolerance and safety of the treatments | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, University Hospital of Nice, Nice, France